CLINICAL TRIAL: NCT04878263
Title: Evaluation and Support Care Process Within the Care Pathway of Heart Failure Patients
Acronym: FIL-EAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: French Cardiology Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-CHITS-04; 2020-A02939-30 (Other: Id-RCB)
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure Acute
Keywords: Acute heart failure; At home hospitalization; Care pathway; Nurse; Geriatric assessment; Social assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Other: Conventional hospitalization
- FIL-EAS ic group (Experimental)
  Interventions: Other: FIL-EAS ic care pathway

INTERVENTIONS:
Other: Conventional hospitalization — Conventional care pathway : patients will be hospitalized as long as necessary and then followed according to High Health Authorities recommendations and usual practices.
  Arms: Control group
Other: FIL-EAS ic care pathway — Organized care pathway with a maximum 4 working day long conventional hospitalization followed by hospitalization at home with a follow up combining hospital and private practice competences.
  Arms: FIL-EAS ic group

SUMMARY:
Acute heart failure current management turns out to be a relative failure considering its elevated economical and human costs and the poor results obtained in terms of disease outcome. Indeed this disease remains associated with a high rate of early re-hospitalizations and low adherence to therapeutic recommended settings and doses. Moreover, extra cardiological follow-up such as in social, geriatric or vaccination fields remain low compared to real needs.

Current recommendations incite health professionals to better define care pathways and to rationalize resources. Guidelines toward creation of hospitalization alternatives or limitation of time spent in hospital are given. In the same time, lack of cardiologic care management within heart failure patient care pathway is associated to poor prognosis and medical desertification as well as resource concentration on important health centers exacerbate this phenomenon. Innovative projects are then needed to improve patient care pathways, to open up areas without specialized health professionals and to rationalize care management by encouraging communication and skill exchange between hospitals and private practices.

FIL-EAS ic projet aims to compare a conventional care pathway in hospital with a follow up defined according to High Authority of Health recommendations to an organized care pathway favoring a short hospitalization (maximum of 4 working days) with early transition, when possible, to a medical and paramedical home care management with an approximately 10 day long combined follow up between hospital and private practices. This second care pathway should help to optimize therapeutics in home living conditions.

DETAILED DESCRIPTION:
Acute heart failure current management turns out to be a relative failure considering its elevated economical and human costs and the poor results obtained in terms of disease outcome. Indeed this disease remains associated with a high rate of early re-hospitalizations and low adherence to therapeutic recommended settings and doses. Current recommendations incite health professionals to better define care pathways and to rationalize resources.

FIL-EAS ic projet aims to compare a conventional care pathway in hospital with a follow up defined according to High Authority of Health recommendations to an organized care pathway favoring a short hospitalization (maximum of 4 working days) with early transition, when possible, to a medical and paramedical home care management with an approximately 10 day long combined follow up between hospital and private practices.

Patients included in the study will be followed up for 6 months with one phone contact one month after hospital discharge, a second one two months later and one consultation 6 months after inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old hospitalized for acute heart failure
* Patient able to express his consent before participating in the study, certified by the caregiver if a written consent is not possible
* Patient able to follow protocol procedures, alone or with a caregiver help
* Caregiver consent to participate in the study and assist the patient during its own participation, if caregiver involvement is necessary
* Patient requiring an hospitalisation of at least 24 hours
* Patient covered by social security or equivalent regimen
* Patient having access to a mobile of fixed phone line

Exclusion Criteria:

* Admission in intensive care or resuscitation unit AND need for inotropic support, vasodilator, or invasive/non-invasive ventilation for the last 24h
* Renal insufficiency with CKD-EPI clearance inferior to 15 ml/min/1.73m2 since admission or dialysis
* Patient planned transfer to a rehabilitation and recuperative care facility (hospital or nursing home)
* Associated disease requiring frequent re-hospitalizations (cancer, dialysis, repeated sessions during planned hospitalizations)
* Associated disease with a high risk of death for the next 6 months
* Chronical respiratory insufficiency requiring daily invasive ventilation or a more than 3L/min permanent oxygen therapy
* Patient suffering from severe dementia defined by a MMSE score ≤ 9
* Person participating in another research testing another care pathway
* Every other reason which, according to investigator, might interfere with study objective assessment
* Person under judicial protection measure (guardianship, curatorship)
* Person deprived of liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
FIL-EAS ic care pathway safety non inferiority | 6 months
  Safety non inferiority will be assessed by comparing the proportion of patients deceased or with unplanned re-hospitalizations for heart failure within the 6 months following randomization between FIL-EAS ic care pathway and conventional hospitalization.

SECONDARY OUTCOMES:
FIL-EAS ic care pathway safety superiority | 6 months
  Safety superiority will be assessed by comparing the proportion of patients deceased or with unplanned re-hospitalizations for heart failure within the 6 months following randomization between FIL-EAS ic care pathway and conventional hospitalization.
Quality of life assessed by EQ-5D questionnaire | 6 months
  Scores obtained after EQ-5D questionnaire completion will be collected during inclusion and research end visit. Evolution between these two scores will be compared between FIL-EAS ic care pathway and conventional hospitalization. EQ-5D questionnaire assess through 5 questions patient mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels : no problems, slight, moderate, severe and finally extreme problems. The patient is asked to tick the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The questionnaire records also patient's self-rated health on a vertical visual analogue scale going from 0 to 100. 0 corresponds to 'The worst health you can imagine' and 100 to 'The best health you can imagine'.
Satisfaction assessed by QSH-37 questionnaire | At the moment of patient initial discharge, up to 3 weeks
  Scores obtained after QSH-37 questionnaire completion will be collected during the visit performed at the end of initial hospitalization and compared between FIL-EAS ic care pathway and conventional hospitalization. The QSH-37 is composed of 37 questions about care management throughout patient hospitalization from the admission until patient's discharge and concerns following elements : relation with professionals (doctors, nurses, housekeepers), response delays, cleanliness, food and room equipment. For each item, possible answers go from "better than desired" to "extremely less than desired".
Cumulative number of days spent in hospital | 6 months
  The cumulative number of days spent in hospital within the 6 months following randomization will be compared between FIL-EAS ic care pathway and conventional hospitalization. In this calculation will be taken into account hospitalizations for acute care, hospitalizations for serious illnesses during their acute phases, mental health activities and non-ambulatory follow-up care and rehabilitation unit stays.
Impact on medical recommendation compliance | 6 months
  Rate of prescription with percentage of recommended dose of heart failure treatments will be collected and compared between the two groups at initial hospitalization discharge and 6 months after. Rate of influenza, pneumococcal and Covid-19 vaccination, percentage of home therapeutic education use, percentage of ambulatory cardiovascular re-education use and rate of acute renal insufficiency occurrence during initial hospitalization will also be assessed.
Geriatric evolution throughout care pathway | 6 months
  Scores obtained at 5 questionnaires will be collected during inclusion visit and research end visit. The evolution of these scores between these two time points will be compared between FIL-EAS ic care pathway and conventional hospitalization. These 5 questionnaires are : ADL (Activities of Daily Leaving), IADL(Instrumental Activities of Daily Leaving)-LAWTON, MNA (Mini Nutritional Assessment), mini GDS (Geriatric Depression Scale) and Dubois 5 words test. The two first asses the ability to perform daily activities. The third one aims at detecting malnutrition cases and is composed of 18 questions. Mini GDS, composed of 4 questions, detects depression cases and finally Dubois 5 words test is a tool evaluating patient cognitive functions. Besides these questionnaires, percentage of geriatric consultation occurrence throughout study participation will be compared between the two care pathways.
Predictive value of biological analyses | 6 months
  Biological analyses results performed throughout study participation will be compared between FIL-EAS ic care pathway and conventional hospitalization and their predictive value with respect to the occurrence of unplanned re-hospitalizations for heart failure or deaths will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Tartière, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (2):
- France (2):
  - Hôpital Sainte Anne, Toulon, Var
  - Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tartiere JM, Candel J, Caignec ML, Jaunay L, Patin C, Kesri-Tartiere L, Esteveny M, Harel M, Derksen H, Quaino G, Lecardonnel I, Challal F, Armangaud P, Birgy C. Assessment of Noninferiority in Terms of 6-month Morbidity and Mortality Rates of a Hospital-at-home Care Pathway for Patients With Acute Heart Failure: FIL-EAS-ic Study Protocol. J Card Fail. 2025 Jun;31(6):928-938. doi: 10.1016/j.cardfail.2024.09.016. Epub 2024 Oct 23. PMID 39454939